CLINICAL TRIAL: NCT06534359
Title: Pilot Trial Comparing Transpyloric to Gastric Feeding in Very Preterm Infants With Bronchopulmonary Dysplasia
Brief Title: Transpyloric Versus Gastric Feeding in Bronchopulmonary Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Erik Allen Jensen, Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-021698
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia; Gastroesophageal Reflux
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Gastroesophageal Reflux | interventions — Enteral Nutrition

STUDY DESIGN:
Masking Description: Randomization procedures will be masked to initial pH-MII testing results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transpyloric tube feeding (Experimental): Nasal or oral placed feeding tube with the distal end located within the second or third portion of the duodenum. Correct placement confirmed by radiograph.
  Interventions: Other: Transpyloric tube feeding
- Gastric tube feeding (Experimental): Nasal or oral placed feeding tube with distal end located within the stomach. Correct placement confirmed by point of care aspirate pH testing or radiograph based on local clinical standard.
  Interventions: Other: Gastric tube feeding

INTERVENTIONS:
Other: Transpyloric tube feeding — Tube feeding into the small bowel
  Arms: Transpyloric tube feeding
Other: Gastric tube feeding — Tube feeding into the stomach
  Arms: Gastric tube feeding

SUMMARY:
The goal of this clinical trial is to learn if transpyloric tube feeding (feeding directly into the small intestine) versus gastric tube feeding tolerably and effectively reduces gastroesophageal reflux in infants born premature who have been diagnosed with bronchopulmonary dysplasia. The main questions this trial aims to answer are:

Does transpyloric as compared to gastric tube feeding result in differences in the amount of experienced hypoxemia (low oxygen level in the blood) or serious adverse events?

Does transpyloric as compared to gastric tube feeding reduce the frequency and severity of gastroesophageal reflux (GER) measured using 24 hour esophageal pH-multichannel intraluminal impedance (pH-MII) monitoring?

Participants will:

Undergo pre-trial 24 hour pH-MII monitoring to determine baseline severity of GER.

Be randomly assigned to receive transpyloric or gastric tube feeding for 2 weeks.

Undergo repeat pH-MII at the end of the 2 week trial to assess for change in GER.

Undergo continuous pulse oximetry to record level of hypoxemia during the 2 week trial.

Undergo saliva and airway (if supported by a breathing tube) fluid collection to measure biomarkers of GER.

Be monitored clinically for possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Birth <32 weeks' gestation
2. Current postmenstrual age of 36-65 weeks
3. Grade 2-3 bronchopulmonary dysplasia (BPD: treatment with positive airway pressure at 36 weeks' PMA) or grade 1 BPD (treatment with ≤2L/min flow nasal cannular at 36 weeks' PMA) with subsequent need for prolonged positive airway pressure and full enteral tube feedings
4. Treatment with positive airway pressure (high flow nasal cannula, non-invasive positive airway pressure, or invasive ventilation) at enrollment

(4) Full gastric tube feedings (≥100mL/kg/d) at the time of enrollment (5) Parental consent to participate

Note: At least 20 infants receiving invasive ventilation will be enrolled to enable endotracheal biomarker testing.

Exclusion Criteria:

1. Transpyloric feedings received within 7d of enrollment
2. Use of a gastric acid suppression, GI promotility drug, or caffeine within 7d of enrollment
3. History of gastrostomy tube placement, gastric fundoplication, or bowel resection resulting in short gut with contraindication to transpyloric feeding
4. Plan to wean off positive airway pressure (for non-intubated subjects) or to be extubated to non-invasive support (for subjects receiving invasive ventilation) within the 2wk trial
5. Known intolerance to transpyloric feeding
6. Persistent >20% endotracheal tube leak (for intubated subjects only)
7. Active treatment with an investigational therapy as part of another interventional trial
8. severe congenital or genetic abnormality that adversely affects GI or cardiopulmonary function

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of time per day with oxygen saturation <80% | During the 2 week trial
  Oxygen saturation will be measured by continuous pulse oximetry throughout the 2 week trial. The proportion of time per day with an oxygen saturation (SpO2) less than 80% will be calculated and reported as a median value observed over the 2 week trial.
Serious adverse events | Until hospital discharge
  A serious adverse event (SAE) will be defined as any adverse experience that is at least possibly related to the study intervention and results in any of the following outcomes:
  * death,
  * a life-threatening event (at risk of death at the time of the event),
  * prolongation of existing hospitalization beyond what would be expected for a preterm infant who requires extended respiratory support near and beyond term corrected gestation, or
  * a persistent or significant disability/incapacity.

SECONDARY OUTCOMES:
Total number of gastroesophageal reflux (GER) episodes | 24 hours
  The total number of GER episodes during a 24 hour period will be measured using 24 hour esophageal pH-multichannel intraluminal impedance (pH-MII) monitoring. Testing is performed by inserting a pH-MII catheter into the esophagus via the nasal or oral route. Reflux episodes are recorded during a 24 hour monitoring period and the total number is tabulated. 24 hour pH-MII testing will be performed prior to randomization and on day 14 (last day) of the clinical trial.
Proportion of GER episodes reaching the proximal pH-MII sensor | 24 hours
  The number of GER episodes detected by 24 hour esophageal pH-MII monitoring that reach the proximal sensor will be recorded and divided by the total number of recorded impedance episodes (regardless of esophageal height)
Total number of pH (acid) only reflux episodes | 24 hours
  The total number of reflux episodes with a pH<4 will be recorded during 24 hour pH-MII monitoring
Salivary and tracheal pepsin concentration | 1 day prior to initiating the trial and on trial day 7 and 14.
  Saliva and tracheal samples will be collected by gentle suctioning and analyzed for concentration of pepsin, a biomarker of GER. Quantification will be performed using commercially available assay.
Salivary and tracheal total bile acid concentration | 1 day prior to initiating the trial and on trial day 7 and 14.
  Saliva and tracheal samples will be collected by gentle suctioning and analyzed for concentration of bile acids, a biomarker of gastro-duodeno reflux. Quantification will be performed using commercially available assay.
Intermittent hypoxemic episodes | During the 2 week trial
  Occurrence of hypoxemic episodes will be recorded using continuous pulse oximetry. Intermittent episodes will be defined as oxygen saturation (SpO2) values <80% lasting longer than 10 seconds.
Prolonged hypoxemic episodes | During the 2 week trial
  Occurrence of hypoxemic episodes will be recorded using continuous pulse oximetry. Prolonged episodes will be defined as oxygen saturation (SpO2) values <80% lasting longer than 60 seconds.
Clinically diagnosed aspiration events | During the 2 week trial
  Aspiration events will be diagnosed as will define aspiration as a witnessed regurgitation (milk in the mouth, clothing respiratory equipment, etc.) event with subsequent clinical decompensation (increase in inspired oxygen by an absolute difference of 20% or more or an increase in delivered mean airway pressure by at least 5cm H2O for ≥ 24 hours beginning within 24 hours of the observed regurgitation event.
Respiratory severity score | During the 2 week trial
  Respiratory severity score is calculated as the delivered mean airway pressure multiplied by supplemental oxygen level. Values will be computed as the daily time weighted average.
Face, Legs, Activity, Cry, Consolability (FLACC) behavioral pain scale | During the 2 week trial
  The FLACC scale assesses pain by observing five categories of behaviors and assigning a score of 0-2 to each category, resulting in a total score of 0-10:
  Face: Facial expressions, such as a smile, grimace, or frown Legs: Leg movement, such as kicking, drawing legs up, or remaining relaxed Activity: Movement, such as lying quietly, squirming, or remaining tense Cry: Crying, moaning, whimpering, or complaining Consolability: Response to comfort, such as being reassured by touching or hugging, or being difficult to console
  FLACC scores will be assessed during routine nursing care (at least twice daily) and summarized as median daily values
Total daily narcotic exposure | During the 2 week trial
  Total dose of narcotic medications received during the 2 week trial will be tabulated in morphine and midazolam equivalents and summarized as mg/kg exposure.
Feeding tube replacement | During the 2 week trial
  Number of times the feeding tube is replaced due to dysfunction or inadvertent dislodgment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania